CLINICAL TRIAL: NCT04304898
Title: An International Patient-led Registry in Fibrotic Interstitial Lung Diseases Using eHealth Technology: I-FILE
Brief Title: An International Patient-led Registry in Fibrotic Interstitial Lung Diseases Using eHealth Technology
Acronym: I-FILE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Principal investigator, Erasmus Medical Center
Other Study IDs: MEC-2020-0029
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Fibrosis
Keywords: eHealth; home spirometry
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Intervention group without a control group
  Interventions: Other: Home spirometry

INTERVENTIONS:
Other: Home spirometry — * Patients will perform daily home spirometry for three months with a Bluetooth-enabled validated, CE-marked home spirometer (Spiro bank Smart, MIR, Italy). Subsequently, patients will perform weekly home spirometry for two years in total. During this period, patients will be asked to perform three measurements each week on the same day.
  * Hospital-based spirometry will be performed according to international guidelines.
  * Patients will complete patient-reported outcomes (PROMs) online in the secured application every six months.

SUMMARY:
The I-FILE study is a prospective multicenter, multinational observational study where the feasibility of a patient-led registry using home monitoring in patients with pulmonary fibrosis will be evaluated. The aim of the study is to gain more insights in disease behavior in patients with pulmonary fibrosis, so in future patients with progressive disease can be better identified.

DETAILED DESCRIPTION:
Nowadays, identifying disease progression will have direct treatment implications in patients with fibrotic Interstitial lung diseases (F-ILDs). eHealth could be a possible solution for close monitoring and detecting disease progression, at a low burden for patients and healthcare providers. The main aim of the I-FILE study will be to evaluate feasibility of a patient-led registry using home spirometry to monitor disease progression in patients with F-ILD. The secondary aim will be to better validate existing health-related quality of life questionnaires to assess the impact of disease and treatment in these patients.

In total 500 patients with newly diagnosed F-ILD will be included. Patients will perform daily home spirometry in the first three months followed by once weekly measurements with a follow up period of 2 years. In addition, patient-reported outcomes (PROMs) will be completed online every 6 months. Results are encrypted and directly sent to a secured server through the online I-FILE application.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed patients with F-ILD according to the ATS/ERS criteria by a multidisciplinary ILD team :

* MDT diagnosis ≤ 6 months before inclusion
* Treatment for F-ILD ≤ than 1 month

Exclusion Criteria:

* Not able to speak, read or write in the native language of the country where the patient is included
* Not able to comply to the study protocol, according to the judgement of the investigator and/or patient
* No access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 untreated patients with a diagnosis of F-ILD in ILD expert centers in 5 European countries
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) home spirometry | 6 months after inclusion
  FVC change measured with home spirometry and saturation at 6 months (in % and L)
Forced Vital Capacity (FVC) home spirometry | 12 months after inclusion
  FVC change measured with home spirometry and saturation at 12 months (in % and L)
Forced Vital Capacity (FVC) home spirometry | 24 months after inclusion
  FVC change measured with home spirometry and saturation at 24 months (in % and L)
Forced Vital Capacity (FVC) hospital spirometry | 6 months after inclusion
  FVC change measured with hospital spirometry and saturation at 6 months (in % and L)
Forced Vital Capacity (FVC) hospital spirometry | 12 months after inclusion
  FVC change measured with hospital spirometry and saturation at 12 months (in % and L)
Forced Vital Capacity (FVC) hospital spirometry | 24 months after inclusion
  FVC change measured with hospital spirometry and saturation at 24 months (in % and L)
Adherence to daily home spirometry | 3 months after inclusion
  The percentage of patients completed daily home spirometry
Adherence to weekly home spirometry | 2 years after inclusion
  The percentage of patients completed weekly home spirometry
L-PF Impacts | Baseline
  • Living with Pulmonary Fibrosis: 21-item questionnaire which assess the way pulmonary fibrosis has impact on quality of life. Total scores range from 0-4, with a higher score indicating more impact of lung fibrosis on the quality of life.
K-BILD | Baseline
  • King's brief Interstitial Lung Disease Health Status: The K-BILD health status questionnaire is a 15 item validated, self-completed heath status questionnaire. It has three domains: breathlessness and activities, psychological and chest symptoms. The K-BILD domain and total score ranges are 0-100, with the higher scores corresponding with better HRQOL. It will take about 3 minutes to complete this questionnaire.
EQ5D | Baseline
  • The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status.
VAS | Baseline
  • Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
LCQ | Baseline
  • Leicester Cough Questionnaire: Cough-specific, health related quality of life is assessed with the Leicester Cough Questionnaire (LCQ), a 19-item questionnaire that has been validated in acute and chronic cough. The overall score ranges from 3 to 21 with a higher score indicating a better quality of life. It will take about 4 minutes to complete the questionnaire.
FAS | Baseline
  • Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
WPAI | Baseline
  • Work Productivity and Activity Impairment Questionnaire: General Health (WPAI) All patients in the working age population will complete this questionnaire which assess loss of work productivity due to disease in six questions .It will take about 2-3 minutes to complete. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
GRoC | Baseline
  • Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
L-PF Impacts | After 12 months
  • Living with Pulmonary Fibrosis: 21-item questionnaire which assess the way pulmonary fibrosis has impact on quality of life. Total scores range from 0-4, with a higher score indicating more impact of lung fibrosis on the quality of life.
K-BILD | After 12 months
  • King's brief Interstitial Lung Disease Health Status: The K-BILD health status questionnaire is a 15 item validated, self-completed heath status questionnaire. It has three domains: breathlessness and activities, psychological and chest symptoms. The K-BILD domain and total score ranges are 0-100, with the higher scores corresponding with better HRQOL. It will take about 3 minutes to complete this questionnaire.
EQ5D | After 12 months
  • The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status.
VAS | After 12 months
  • Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
LCQ | After 12 months
  • Leicester Cough Questionnaire: Cough-specific, health related quality of life is assessed with the Leicester Cough Questionnaire (LCQ), a 19-item questionnaire that has been validated in acute and chronic cough. The overall score ranges from 3 to 21 with a higher score indicating a better quality of life. It will take about 4 minutes to complete the questionnaire.
FAS | After 12 months
  • Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
WPAI | After 12 months
  • Work Productivity and Activity Impairment Questionnaire: General Health (WPAI) All patients in the working age population will complete this questionnaire which assess loss of work productivity due to disease in six questions .It will take about 2-3 minutes to complete. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
GRoC | After 12 months
  • Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
L-PF Impacts | After 24 months
  • Living with Pulmonary Fibrosis: 21-item questionnaire which assess the way pulmonary fibrosis has impact on quality of life. Total scores range from 0-4, with a higher score indicating more impact of lung fibrosis on the quality of life.
K-BILD | After 24 months
  • King's brief Interstitial Lung Disease Health Status: The K-BILD health status questionnaire is a 15 item validated, self-completed heath status questionnaire. It has three domains: breathlessness and activities, psychological and chest symptoms. The K-BILD domain and total score ranges are 0-100, with the higher scores corresponding with better HRQOL. It will take about 3 minutes to complete this questionnaire.
EQ5D | After 24 months
  • The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status.
VAS | After 24 months
  • Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
LCQ | After 24 months
  • Leicester Cough Questionnaire: Cough-specific, health related quality of life is assessed with the Leicester Cough Questionnaire (LCQ), a 19-item questionnaire that has been validated in acute and chronic cough. The overall score ranges from 3 to 21 with a higher score indicating a better quality of life. It will take about 4 minutes to complete the questionnaire.
FAS | After 24 months
  • Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
WPAI | After 24 months
  • Work Productivity and Activity Impairment Questionnaire: General Health (WPAI) All patients in the working age population will complete this questionnaire which assess loss of work productivity due to disease in six questions .It will take about 2-3 minutes to complete. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
GRoC | After 24 months
  • Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
Time to change of L-PF Impacts | 2 years
  • Living with Pulmonary Fibrosis: 21-item questionnaire which assess the way pulmonary fibrosis has impact on quality of life. Total scores range from 0-4, with a higher score indicating more impact of lung fibrosis on the quality of life.
Time to change of K-BILD | 2 years
  • King's brief Interstitial Lung Disease Health Status: The K-BILD health status questionnaire is a 15 item validated, self-completed heath status questionnaire. It has three domains: breathlessness and activities, psychological and chest symptoms. The K-BILD domain and total score ranges are 0-100, with the higher scores corresponding with better HRQOL. It will take about 3 minutes to complete this questionnaire.
Time to change of EQ5D | 2 years
  • The EuroQol five dimensions 5-level questionnaire: 6-item questionnaire on five dimensions: The EuroQol five dimensions 5-level questionnaire is a standardized instrument to measures health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher score indicates a poorer health status.
Time to change of VAS | 2 years
  • Visual Analogue Scale: scores on fatigue, dyspnea, cough and general wellbeing on a scale ranging from 0-10. Higher score indicates more complaint.
Time to change of LCQ | 2 years
  • Leicester Cough Questionnaire: Cough-specific, health related quality of life is assessed with the Leicester Cough Questionnaire (LCQ), a 19-item questionnaire that has been validated in acute and chronic cough. The overall score ranges from 3 to 21 with a higher score indicating a better quality of life. It will take about 4 minutes to complete the questionnaire.
Time to change of FAS | 2 years
  • Fatigue Assessment Scale: 10-item questionnaire about fatigue FAS. The fatigue assessment scale (FAS) is a 10-item self-administered questionnaire about fatigue in patients with sarcoidosis. The score ranges from 5-50 points, with a score of ≥ 22 points as cut-off for fatigue. The minimal important difference (MID) is 4 points or a 10% lower score. It will take about 1-2 minutes to complete.
Time to change of WPAI | 2 years
  • Work Productivity and Activity Impairment Questionnaire: General Health (WPAI) All patients in the working age population will complete this questionnaire which assess loss of work productivity due to disease in six questions .It will take about 2-3 minutes to complete. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time to change of GRoC | 2 years
  • Global Rating of Change Scales: Global rating of change (GRC) scales provide a method of obtaining information about improving or deteriorated of health condition of patients over time. Patients are asked to make global ratings on changes in regards to their well-being on a 15-point self-report scale (from -7 to 7 ). It will take about 1 minute to complete. Higher score indicates a better health condition.
Predictors | 2 years
  Predictors of disease progression and mortality
FVC change hospital-based and home spirometry | 2 years
  Correlations between FVC change between home and hospital-based spirometry
FVC change and HRQOL and symptom changes | 12 months
  Correlations between FVC change and HRQOL and symptom changes
FVC change and HRQOL and symptom changes | 24 months
  Correlations between FVC change and HRQOL and symptom changes
Differences in adherence between countries | 2 years
  Differences in adherence, FVC change, HRQOL and mortality between countries
Healthcare provider and patient satisfaction | 2 years
  Healthcare provider and patient satisfaction and experience with the online application. Patients and healthcare providers are asked about their experiences and opinions on homemonitoring.
Mortality | 2 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Wijsenbeek, MD PhD, Principal Investigator — Erasmus Medical Center; Wim Wuyts, MD PhD, Principal Investigator — Universitair Ziekenhuis Leuven; Anna-Maria Hoffmann-Vold, MD PhD, Principal Investigator — Oslo University Hospital; Michael Kreuter, MD PhD, Principal Investigator — Interdisciplinary Center for Sarcoidosis, Thoraxklinik, University Hospital Heidelberg; Philip Molyneaux, MD PhD, Principal Investigator — Royal Brompton Hospital, Guys and St Thomas' Hospital NHS Foundation Trust.; Vincent Cottin, MD PhD, Principal Investigator — Service de pneumologie, hôpital Louis Pradel, Hospices Civils de Lyon; Katarina Antoniou, Principal Investigator — Laboratory of Molecular and Cellular Pneumonology, Respiratory Medicine Department, School of Medicine, University of Crete, Heraklion, Greece
Locations (2):
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nakshbandi G, Moor CC, Antoniou K, Cottin V, Hoffmann-Vold AM, Koemans EA, Kreuter M, Molyneaux PL, Wuyts WA, Wijsenbeek MS. Study protocol of an international patient-led registry in patients with pulmonary fibrosis using online home monitoring: I-FILE. BMC Pulm Med. 2023 Feb 2;23(1):51. doi: 10.1186/s12890-023-02336-4. PMID 36732734